CLINICAL TRIAL: NCT01279954
Title: An Openlabel, Phase II Trial of Abatacept (Orencia) in the Treatment of Refractory Non-infectious Uveitis.
Brief Title: Abatacept in the Treatment of Uveitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Eric B. Suhler, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: e7035
Record Dates: First submitted 2011-01-14; First posted 2011-01-20 (Estimated); Results first posted 2019-02-21 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-01

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis | interventions — Abatacept

ARMS (2):
- open-label abatacept first, then 5 mg/kg abatacept (Experimental): 10 mg/kg abatacept (6 months). Then 5 mg/kg abatacept (18 months)
  Interventions: Drug: Abatacept
- open-label abatacept first, then 10 mg/kg abatacept (Experimental): 10 mg/kg abatacept (6 months). Then 10 mg/kg abatacept (18 months)
  Interventions: Drug: Abatacept

INTERVENTIONS:
Drug: Abatacept — Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then be randomized to receive either 5 mg/kg or 10 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
  Other Names: orencia

SUMMARY:
The purpose of this study is to assess the safety and efficacy of abatacept in the treatment of uveitis.

ELIGIBILITY:
Inclusion Criteria:

* patients with vision-threatening autoimmune uveitis
* failure to respond to prednisone and at least one other systemic immunosuppressive, or intolerance to such medications due to side effects

Exclusion Criteria:

* serious concomitant illness that could interfere with the subject's participation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric B. Suhler, MD, MPH, Principal Investigator — Oregon Health and Science University; James T Rosenbaum, MD, Study Director — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Abatacept, Then 10 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then 10 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- Open-label Abatacept, Then 5mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then 5 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
Period: Overall Study
Arm/Group | Open-label Abatacept, Then 10 mg/kg Abatacept | Open-label Abatacept, Then 5mg/kg Abatacept
Started | 5 | 5
Completed | 2 | 1
Not Completed | 3 | 4
Not completed — Lack of Efficacy | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Open-label Abatacept, Then 5 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then 5 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- Total: Total of all reporting groups
Arm/Group | Open-label Abatacept, Then 10 mg/kg Abatacept | Open-label Abatacept, Then 5 mg/kg Abatacept | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 1 | 3
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10
Ocular Inflammation [Count of Participants; unit: Participants] — Ocular inflammation present at baseline, judged by fluorescein angiography, vitreous haze, and/or anterior chamber inflammation.
  Participants | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: number of participants with adverse events
Time Frame: 2 years
Population: 2 subjects were randomized to the 5 mg/kg abatacept group but one of these subjects only received 1 treatment before being removed from the study due to worsening. Only 1 of the 2 subjects randomized to this group completed the study. This explains the discrepancy between this table and the participant flow.
Measure: Count of Participants; unit: Participants
Groups:
- Randomized 10 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then continue receiving 10 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- Randomized 5 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then receive 5 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- Open Label Abatacept: All subjects received open label 10mg/kg abatacept during the first 24 weeks of the trial.
Arm/Group | Randomized 10 mg/kg Abatacept | Randomized 5 mg/kg Abatacept | Open Label Abatacept
Number analyzed (Participants) | 2 | 2 | 10
Participants | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Improvement by 2 or More Lines of Best-corrected Visual Acuity
Description: improvement by 2 or more lines of best-corrected visual acuity With the outcome measure being at 24 weeks, only one group is analyzed. All the subjects received open-label abatacept at 10 mg/kg during the first 24 weeks.
Time Frame: Week 24
Population: All subjects started the trial on open label abatacept, so only one group is being analyzed for this 24 week outcome.
Measure: Count of Participants; unit: Participants
Groups:
- Open-label Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then be randomized to receive either 5 mg/kg or 10 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 10
Participants | 0

3. Secondary Outcome: Number of Participants With Reduction in Systemic Corticosteroid or Other Immunosuppressive Therapy by at Least 50%
Description: Reduction in dose of systemic corticosteroid or other immunosuppressive therapy by at least 50% With the outcome measure being at 24 weeks, only one group is analyzed. All the subjects received open-label abatacept at 10 mg/kg during the first 24 weeks.
Time Frame: Week 24
Population: With the outcome measure being at 24 weeks, only one group is analyzed. All 10 subjects received open-label abatacept at 10 mg/kg during the first 24 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 8
Participants | 6

4. Secondary Outcome: Number of Participants With Control of Ocular Inflammation, as Judged on Clinical Criteria, According to Standard Methods
Description: Reduction of AC cellular activity and/or vitreous haze by 2 grades. Reduction of chorioretinal infiltrates or reduction of retinal vasculitis. Reduction of cystoid macular edema and/or retinal inflammation. With the outcome measure being at 24 weeks, only one group is analyzed. All the subjects received open-label abatacept at 10 mg/kg during the first 24 weeks.
Time Frame: Week 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Open-label Abatacept
Number analyzed (Participants) | 9
Participants | 4

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- 10 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then receive 10 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- 5 mg/kg Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial. At 6 months subjects will then receive 5 mg/kg.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
- Open Label Abatacept: Abatacept: Subjects will receive approximately 10 mg/kg rounded to the nearest 25 mg for the first 6 months of the trial.
  Abatacept will be administered as a 30-minute intravenous infusion. Following the initial administration, abatacept will be given at 2 and 4 weeks after the first infusion and every 4 weeks thereafter for up to 2 years.
Arm/Group | 10 mg/kg Abatacept | 5 mg/kg Abatacept | Open Label Abatacept
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/10
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT01279954/Prot_SAP_000.pdf